CLINICAL TRIAL: NCT01347138
Title: Health Care Management for the Elderly in Community Through Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Clinical Research Coordination Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Hyeon Woo Yim, Professor, National Clinical Research Coordination Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: A102065
Record Dates: First submitted 2011-04-27; First posted 2011-05-04 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Major Depressive Disorders; Senile; Depression
Keywords: Screening; depression; case management
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- case management (Experimental): case management regulary
  Interventions: Other: case management
- Control (No Intervention): usual care

INTERVENTIONS:
Other: case management — confirmation of hospital visit date, checking the adverse effect and treatment compliance
  Arms: case management

SUMMARY:
Depression in late life has been associated with losses in functioning and quality of life, mortality, and increased health care costs. Although late life depression can be successfully treated with antidepressant medication or psychotherapy, few older adults receive adequate trials of such treatment in community in Korea. Barriers, such as loss of loved ones, medical illnesses, and social stigma associated with depression, lack of social and financial support, to effective treatment of depression can be especially problematic for older adult. Screening has been valuable in overcoming barriers to diagnosis. Over 60 year old community dwelling people will be screened for symptoms of four geriatric conditions (depression, dementia, urinary incontinence, and sleep disorder). Those who will be screened positive for each condition will be refer to clinic for diagnosis. Among them only those cases confirmed as depression by psychiatrists will be enrolled in this study. Enrolled patients will be randomly assigned to either case management or usual care conditions.

The objective of the study is to test whether a system of screening, assessment, and follow-up provided by case manager improves in recognizing the target geriatric conditions (depression, dementia, urinary incontinence, and sleep disorder) and healthcare outcomes.

ELIGIBILITY:
Inclusion Criteria:

* over 60 year old
* having medicare insurance

Exclusion Criteria:

* dementia and other psychiatric disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Geriatric Depression Score | 6 months after baseline

SECONDARY OUTCOMES:
quality of life | 6 months after baseline
treatment compliance | 6 months after baseline
suicide ideation | 6 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon Woo Yim, MD. Ph.D., Principal Investigator — The Catholic University of Korea
Locations (1):
- City of Choongju public health center, Choongju, Choongchungbuk-Do, South Korea